CLINICAL TRIAL: NCT04238182
Title: Short Term Effect of Wet Versus Dry Cupping on Chest Expansion in Sedentary Smokers
Brief Title: Short Term Effect of Interscapular Cupping on Chest Expansion in Sedentary Male Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/002576
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wet cupping (Active Comparator): smokers in this group will receive single wet cupping session
  Interventions: Other: wet cupping
- dry cupping (Active Comparator): smokers in this group will receive single dry cupping session
  Interventions: Other: dry cupping

INTERVENTIONS:
Other: wet cupping — This smoker group will receive single wet cupping session. The first site is between the two scapulae (interscapular), opposite the T1-T3 scapular spine. This area is called Al-Kahil in Arabic. The second site is located on the spinous process of seventh cervical vertebra and it is called GV14 in Chinese medicine. The third site is BL-17 (Ge Shu Diaphragm Shu) is located 1.5 cun lateral to the lower border of the spinous process of the seventh thoracic vertebra (T7). BL 17 can directly act on the septum transversum of diaphragm . Cupping of BL 17 will be done bilaterally.
  Arms: wet cupping
Other: dry cupping — The smoker group will receive single dry cupping session. The first site is between the two scapulae (interscapular), opposite the T1-T3 scapular spine. This area is called Al-Kahil in Arabic. The second site is located on the spinous process of seventh cervical vertebra and it is called GV14 in Chinese medicine. The third site is BL-17 (Ge Shu Diaphragm Shu) is located 1.5 cun lateral to the lower border of the spinous process of the seventh thoracic vertebra (T7). BL 17 can directly act on the septum transversum of diaphragm. Cupping of BL 17 will be done bilaterally.
  Arms: dry cupping

SUMMARY:
Although cupping remains a popular treatment modality worldwide, its efficacy for most health issues has not been scientifically evaluated so further studies are needed . Claims of cardiac, vascular and respiratory protective role of inter-scapular (alkhil cupping). No studies investigated the acute effect of wet versus dry cupping - on an important cupping area like alkhil hence the importance of this study comes.

DETAILED DESCRIPTION:
The interscapular area is used for wet cupping therapy (WCT) and was found to have special features: brown adipose tissue, immediate proximity to sympathetic ganglia, passage of the thoracic duct, two important acupuncture meridians, and proximity to the main vessel divisions carrying blood from the heart and the brain. These features indicate that the interscapular application of WCT not only discharges waste materials through a shifting of blood to the site after application of a traction force but also invigorates the body's metabolism, increases immunity, and regulates blood biochemistry, which are desired therapeutic effects of WCT.

One of known in Sunnah and in Arabic main cupping points of interscapular area is (alkahil), opposite to thoracic (T) T1-T3 scapular spine .

Prophetic medicine was our reference in selecting back points e.g. the Kahel region seems to be the most suitable point for practicing Al-hijamah for therapeutic and preventive purposes and is regarded as a common place for clearing blood coming to the skin circulation in treating many disease conditions. Kahel region is a prominent anatomical landmark and its surface marking is easy to be detected on the midline of the back at the junction of the back of the neck with the back region. Other related positions can be defined as above kahel region, below kahel region, to the right of kahel region and to the left of it.

Prophetic medicine recommended to practice Alhijamah on mainly skin over 7th cervical (C7) vertebral spine to get the maximal therapeutic benefit. Gavernorer vessel (GV) GV 14, one of the cardinal points of the governing channel, is also located next to the interscapular site on or just below the spinous process of C7. Unblocking this point, which is associated with general energy excess, may balance the functions of all body organs. Clearly, more investigations are needed to clarify every facet of activating the functions of GV cardinal points during WCT applied to the interscapular area.

Before starting the study, clearance will be obtained from the institutional ethical committee and prior informed consent of all the participants will be obtained before conducting the study.

forty smoker men will be randomly selected and divided to 2 groups equal in number for each. (Group A) will receive single wet cupping session. (Group B) will receive single dry cupping session. The following points will be selected for cupping in both groups. The first site is between the two scapulae (interscapular), opposite the T1-T3 scapular spine. This area is called Al-Kahil in Arabic. The second site is located on the spinous process of seventh cervical vertebra and it is called GV14 in Chinese medicine. The third site is BL-17 (Ge Shu Diaphragm Shu) is located 1.5 cun lateral to the lower border of the spinous process of the seventh thoracic vertebra (T7). BL 17 can directly act on the septum transversum of diaphragm. Cupping of bladder 17 will be done bilaterally.

ELIGIBILITY:
Inclusion Criteria:

1. 40 healthy sedentary male smokers.
2. Body mass index of participants will range between < 30 kg/m².
3. The volunteers will have no record of any cupping type, and/or other complementary and treatments in the previous 6 months.
4. The volunteers with no specific causes of stress.

Exclusion Criteria:

1. Alcoholic and addicted volunteers.
2. Current use of anticoagulants and /or coagulopathy.
3. History of chronic or acute pulmonary and cardiac diseases
4. Congenital or acquired chest wall deformities.
5. Apparent or any history of chest trauma

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-02-07 (Estimated); Study Completion 2020-02-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | immediately after the session
  - Sitting position is usually adequate for routine measurement of blood pressure, participants will be in sitting position with back supported for 5 minutes, with arm bared , supported at the level of the heart as (denoted by the mid-sternal level), in quiet warm setting is required, no caffeine for preceding 30 minutes, question about the most recent meal or evacuation of bowels or bladder. Distended abdominal viscera cause blood pressure elevation presumably because of anxiety.
oxygen saturation | immediately after the session
  by pulse oximeter

SECONDARY OUTCOMES:
heart rate | immediately after the session
  by pulse oximeter
chest expansion | immediately after the session
  - The chest expansion will be taken as thoracic circumference at the end of forced inspiration minus thoracic circumference at the end of forced expiration. Two readings from upper and lower thoracic expansion will be measured at an interval of 5 minutes with the inelastic tape around the body. The averages of the two readings will be recorded. For the upper thoracic excursion (UCE), the tape measure will be placed at the level of the fifth thoracic spinous process and the third intercostal space at the midclavicular line and for the lower thoracic excursion (LCE), the tape measure will be placed at the level of the 10th thoracic spinous process and the tip of the xiphoid process. Measurements will be taken at the height of maximal inspiration and expiration and considerable care will be exercised not to pull the tape too tightly while making the measurements

CONTACTS AND LOCATIONS:
Overall Officials: ali ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt